CLINICAL TRIAL: NCT04200352
Title: An Open-Label, Long-Term Safety, Tolerability, and Efficacy Study of TEV-50717 (Deutetrabenazine) for the Treatment of Dyskinesia in Cerebral Palsy in Children and Adolescents (Open RECLAIM-DCP)
Brief Title: A Study to Test if TEV-50717 is Safe and Effective in Relieving Abnormal Involuntary Movements in Cerebral Palsy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Failure of TV50717-CNS-30080 (parent study) to meet the primary efficacy endpoint
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TV50717-CNS-30081; 2019-001807-19 (EudraCT Number)
Record Dates: First submitted 2019-12-12; First posted 2019-12-16 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy, Dyskinetic
MeSH Terms: conditions — Cerebral Palsy | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TEV-50717 (Experimental): The dose of the TEV-50717 should be increased on a weekly basis to reach a clinically meaningful reduction in dyskinesia, as indicated by a reduction in the Clinical Global Impression of Improvement;(CGI-I).
  Interventions: Drug: TEV-50717

INTERVENTIONS:
Drug: TEV-50717 — Oral tablets are 6, 9, and 12 mg.
  Other Names: Deutetrabenazine, SD-809

SUMMARY:
Study TV50717-CNS-30081 is a 55-week study in which participants who have successfully completed the parent study (Study TV50717-CNS-30080) may be eligible to enroll in this study.

The primary objective of this study is to evaluate the safety and tolerability of long-term therapy with TEV-50717 in children and adolescents with DCP.

The secondary objective of this study is to evaluate the efficacy of long-term therapy with TEV-50717 in reducing the severity of DCP.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed parent Study TV50717-CNS-30080.
* Participant weighs at least 12 kg (26 lb) on day 1 of this study.
* Participant is able to swallow TEV-50717 whole. NOTE- Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Participant has clinically significant depression at screening or day 1 of this study. Note: Participants receiving antidepressant therapy may be enrolled if on a stable dose for at least 6 weeks before screening or day 1 (whichever comes first) and anticipated to remain stable (dose and frequency) within the study duration.
* Participant has a history of suicidal intent or related behaviors based on medical or psychiatric history or the C-SSRS at screening visit, if performed, or at the day 1 visit, as applicable according to the participant's age:

  * intent to act on suicidal ideation with a specific plan, irrespective of level of ambivalence, at the time of suicidal thought
  * suicidal preparatory acts or behavior.
* Participant has a history of a previous actual, interrupted, or aborted suicide attempt.
* Participant has a first-degree relative who has completed suicide.
* Participant has received any of the following concomitant Participant has received any of the following concomitant medications within the specified exclusionary windows from screening or day 1 (whichever comes first) of this study:

  * within 30 days: tetrabenazine or valbenazine
  * within 21 days: reserpine
  * within 14 days: levodopa, dopamine agonists, and monoamine oxidase inhibitors
* Participant has received treatment with stem cells, deep brain stimulation, transmagnetic stimulation, or transcranial direct current stimulation for treatment of abnormal movements or CP since the week 15 visit of Study TV50717-CNS-30080, or the participant is not in a stable clinical condition.
* Participants with a history of torsade de pointes, congenital long QT syndrome, bradyarrhythmias, other cardiac arrhythmias, or uncompensated heart failure.
* Participant has a known allergy to any of the components of TEV-50717.
* Participant has participated in an investigational drug or device study other than Study TV50717-CNS-30080 and received IMP/intervention within 30 days or 5 drug half-lives of day 1 of this study, whichever is longer.
* Participant is pregnant or breastfeeding. NOTE- Additional criteria apply, please contact the investigator for more information

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (30):
- United States (5):
  - Teva Investigational Site 14137, Birmingham, Alabama
  - Teva Investigational Site 14295, San Diego, California
  - Teva Investigational Site 14122, Voorhees Township, New Jersey
  - Teva Investigational Site 14299, Charleston, South Carolina
  - Teva Investigational Site 14129, Nashville, Tennessee
- Teva Investigational Site 39058, Blegdamsvej 9, Denmark
- Israel (2):
  - Teva Investigational Site 80146, Tel-Aviv, Tel-Aviv District
  - Teva Investigational Site 80147, Zerifin, Central District
- Italy (2):
  - Teva Investigational Site 30214, Milan
  - Teva Investigational Site 30216, Pisa
- Poland (4):
  - Teva Investigational Site 53434, Gdansk
  - Teva Investigational Site 53428, Gdansk, Pomerania Province
  - Teva Investigational Site 53427, Krakow
  - Teva Investigational Site 53430, Wiazowna, Mazovia Province
- Russia (8):
  - Teva Investigational Site 50477, Kazan'
  - Teva Investigational Site 50475, Khabarovsk, Khabarovsk Krai Region
  - Teva Investigational Site 50470, Moscow, Moscow Region
  - Teva Investigational Site 50485, Nizhniy Novgorod, Nizhny Novgorod Region
  - Teva Investigational Site 50468, Novosibirsk, Novosibirsk Region
  - Teva Investigational Site 50469, Smolensk, Smolensk Region
  - Teva Investigational Site 50478, Stavropol, Stavropol Krai Region
  - Teva Investigational Site 50474, Tyumen, Tyumen Region
- Teva Investigational Site 31254, Valencia, Spain
- Ukraine (4):
  - Teva Investigational Site 58313, Dnipro, Dnipropetrovsk Province
  - Teva Investigational Site 58309, Kyiv, Kyiv Province
  - Teva Investigational Site 58311, Odessa, Odessa Province
  - Teva Investigational Site 58310, Vinnytsya, Vinnytsia Province
- United Kingdom (3):
  - Teva Investigational Site 34245, Edinburgh, Edinburgh
  - Teva Investigational Site 34243, London, Greater London
  - Teva Investigational Site 34244, Sheffield, South Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 44 participants with dyskinesia in cerebral palsy (DCP) from Study TV50717-CNS-30080 (NCT03813238) rolled over into Study TV50717-CNS-30081.
Groups:
- TEV-50717: TEV-50717 was administered as oral tablets once daily for up to 53 weeks (7 weeks dose titration and 46 weeks maintenance). From Week 1 through Week 7, the dose of TEV-50717 was adjusted according to the titrations scheme (based on body weight and cytochrome P450 2D6 [CYP2D6] impairment status at baseline) to identify a dose level that optimally reduced dyskinesia (as determined by the investigator, as indicated by a reduction in the clinical global impression of improvement [CGI-I]) and was well tolerated. After titration, participants continued to receive their maintenance dose over the next 46 weeks.
Period: Overall Study
Arm/Group | TEV-50717
Started | 44
Received at Least 1 Dose of Study Drug | 44
Completed | 24
Not Completed | 20
Not completed — Death | 1
Not completed — Adverse Event | 6
Not completed — Withdrawal by parent/guardian | 6
Not completed — Lack of Efficacy | 1
Not completed — Other than specified | 6

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717.
Groups:
- TEV-50717: TEV-50717 was administered as oral tablets once daily for up to 53 weeks (7 weeks dose titration and 46 weeks maintenance). From Week 1 through Week 7, the dose of TEV-50717 was adjusted according to the titrations scheme (based on body weight and CYP2D6 impairment status at baseline) to identify a dose level that optimally reduced dyskinesia (as determined by the investigator, as indicated by a reduction in the CGI-I) and was well tolerated. After titration, participants continued to receive their maintenance dose over the next 46 weeks.
Arm/Group | TEV-50717
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.1 (3.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 42
  More than one race | 0
  Unknown or Not Reported | 2
Extrapyramidal Symptom Rating Scale (ESRS) Subscale I Total Score [Mean (Standard Deviation); unit: units on a scale] — ESRS subscale I is a 7-item subjective questionnaire to evaluate parkinsonism, akathisia, dystonia, and dyskinesia. ESRS I is scored on 4-point scale (0=absent, 1=Mild, 2=Moderate, 3=Severe) for each item. The evaluation takes into account the verbal report of participant on 1) frequency and duration of symptom during the day, 2) number of days the symptom was present during the last week, and 3) subjective evaluation of intensity of symptom by the participant. Total score was the sum of 7 items ranging from 0 (absent) to 21 (severe). Higher scores indicate greater severity of disorder.
  units on a scale | 9.7 (3.94)
ESRS Subscale II Total Score [Mean (Standard Deviation); unit: units on a scale] — The ESRS subscale II is a 17-item questionnaire to evaluate parkinsonism and akathisia. The ESRS II consists of the following parts: tremor (0 [none]-48 [severe]), gait and posture (0 [none]-6 [severe]), postural stability (0 [none]-6 [severe]), rigidity (0 [none]-24 [severe]), expressive automatic movements (0 [none]-6 [severe]), bradykinesia (0 [none]-6 [severe]), and akathisia (0 [none]-6 [severe]). Total score was the sum of the 17 items ranging from 0 (absent) to 102 (severe). Higher scores indicate greater severity of disorder.
  units on a scale | 20.7 (19.73)
Child Behavior Checklist (CBCL) Competence Total Score [Mean (Standard Deviation); unit: units on a scale] — CBCL Competence Scale (Parts I to VII) assesses various activities (for example, sports, hobbies, games, organizations, clubs, teams, groups, jobs, and chores), interpersonal relationships, and academic performance. The checklists having 120 questions consist of a number of statements about child's behavior and responses which are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. CBCL competence total score ranged from 0 (no problem) to 240 (greater problem). Higher scores indicate greater problems in child behavior. Population: Here, 'overall number of participants analyzed' = participants evaluable for this Baseline measure.
  units on a scale
    number analyzed (Participants) | 33
    (all) | 11.70 (4.392)
CBCL Syndrome Total Score [Mean (Standard Deviation); unit: units on a scale] — CBCL Syndrome Scale comprises 113 questions related to problem behaviors. For each item, responses are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. Problem behaviors are scored on the following 8 empirically based syndromes: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior. CBCL syndrome total score ranged from 0 (no problem) to 226 (lesser problem). Higher scores indicate greater problems in child behavior.
  units on a scale | 30.7 (21.06)
Epworth Sleepiness Scale (ESS) Total Score [Mean (Standard Deviation); unit: units on a scale] — ESS is a self-administered questionnaire composed of 8 questions that provide a measure of a participant's general level of daytime sleepiness. Responders were asked to rate their chances of falling asleep while engaged at 8 different activities, on a 4-point scale: 0 = would never fall asleep; 1=slight chance of falling asleep; 2=moderate chance of falling asleep; 3=high chance of falling asleep. Total score was calculated as the sum of 8 item scores ranging from 0 (never) to 24 (high chance of falling asleep). Higher scores indicate high chances of falling asleep.
  units on a scale | 2.0 (2.79)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse events can include any of the following: clinically significant vital signs, ECG parameters, or laboratory parameters. An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. SAEs included death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to Week 55
Population: The ITT analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-50717
Number analyzed (Participants) | 44
Participants | 39

2. Primary Outcome: Number of Participants (Aged ≥12 Years) With Columbia-Suicide Severity Rating Scale (C-SSRS) Outcomes (Worst Overall Finding)
Description: Participants were placed into categories for suicidal ideation or behavior and non-suicidal self-injurious behavior based on their responses to various questions. For suicidal ideation or behavior, the following categories were used: None; Wish to be dead; Non-specific active suicidal thoughts; Any methods (not plan) without intent to act; Some intent to act, without specific plan; Specific plan and intent; Preparatory acts or behavior; Aborted attempt; Interrupted attempt; Actual attempt; and Suicide. For non-suicidal self-injurious behavior, the following categories were used: No or yes. Number of participants with worst overall finding of suicidal ideation or suicidal behavior and non-suicidal self-injurious behavior from Baseline to Week 54 are reported.
Time Frame: Baseline to Week 54
Population: The ITT analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717. Here, 'overall number of participants analyzed' = participants who provided a baseline value and at least one post-baseline value for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | TEV-50717
Number analyzed (Participants) | 18
Participants
  Suicidal ideation/behavior - None | 18
  Suicidal ideation/behavior - Wish to be dead | 0
  Suicidal ideation/behavior - Non-specific active suicidal thoughts | 0
  Suicidal ideation/behavior - Any methods (not plan) without intent to act | 0
  Suicidal ideation/behavior - Some intent to act, without specific plan | 0
  Suicidal ideation/behavior - Specific plan and intent | 0
  Suicidal ideation/behavior - Preparatory acts or behavior | 0
  Suicidal ideation/behavior - Aborted attempt | 0
  Suicidal ideation/behavior - Interrupted attempt | 0
  Suicidal ideation/behavior - Actual attempt | 0
  Suicidal ideation/behavior - Suicide | 0
  Non-suicidal self-injurious behavior - No | 18
  Non-suicidal self-injurious behavior - Yes | 0

3. Primary Outcome: Change From Baseline in Extrapyramidal Symptom Rating Scale (ESRS) Subscale I Total Score at Week 54
Description: The ESRS subscale I is a 7-item subjective questionnaire to evaluate parkinsonism, akathisia, dystonia and dyskinesia. The ESRS I is scored on a 4-point scale (0=absent, 1=Mild, 2=Moderate, 3=Severe) for each item. The evaluation takes into account the verbal report of the participant on 1) the frequency and duration of the symptom during the day, 2) the number of days the symptom was present during the last week, and 3) the subjective evaluation of the intensity of the symptom by the participant. Total score was the sum of the 7 items which ranges from 0 (absent) to 28 (severe). Higher scores indicate greater severity of disorder.
Time Frame: Baseline, Week 54
Population: The ITT analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 24
units on a scale | -1.4 (2.02)

4. Primary Outcome: Change From Baseline in ESRS Subscale II Total Score at Week 54
Description: The ESRS subscale II is a 17-item questionnaire to evaluate parkinsonism and akathisia. The ESRS II consists of the following parts: tremor (0 [none]-48 [severe]), gait and posture (0 [none]-6 [severe]), postural stability (0 [none]-6 [severe]), rigidity (0 [none]-24 [severe]), expressive automatic movements (0 [none]-6 [severe]), bradykinesia (0 [none]-6 [severe]), and akathisia (0 [none]-6 [severe]). Total score was the sum of the 17 items ranging from 0 (absent) to 102 (severe). Higher scores indicate greater severity of disorder.
Time Frame: Baseline, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 24
units on a scale | -1.5 (6.41)

5. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Competence Total Score at Week 53
Description: The CBCL assesses behavioral and emotional status in children ages 6 through 18 years of age as reported by the caregiver. The full CBCL has two parts, a Competence Scale (Parts I to VII) and a Syndrome Scale (behavioral items). The Competence Scale (Parts I to VII) assesses various activities (for example, sports, hobbies, games, organizations, clubs, teams, groups, jobs, and chores), interpersonal relationships, and academic performance. The checklists having 120 questions consist of a number of statements about the child's behavior and responses which are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. CBCL competence total score ranged from 0 (no problem) to 240 (lesser problem), which was calculated by adding individual scores of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 20
units on a scale | 0.49 (3.018)

6. Primary Outcome: Change From Baseline in CBCL Syndrome Total Score at Week 53
Description: The CBCL assesses behavioral and emotional status in children ages 6 through 18 years of age as reported by the caregiver. The full CBCL has two parts, a Competence Scale (Parts I to VII) and a Syndrome Scale (behavioral items). The Syndrome Scale comprises 113 questions related to problem behaviors. For each item, the responses are recorded on a scale: 0 = Not True; 1 = Somewhat or Sometimes True; 2 = Very True or Often True. The problem behaviors are scored on the following 8 empirically based syndromes: anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior, and aggressive behavior. CBCL syndrome total score ranged from 0 (no problem) to 226 (lesser problem), which was calculated by adding individual scores of each domain. Higher scores indicate greater problems in child behavior.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 25
units on a scale | -1.7 (14.96)

7. Primary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Week 54
Description: The ESS is a self-administered questionnaire composed of 8 questions that provide a measure of a participant's general level of daytime sleepiness. The ESS is composed of 8 items. The responders were asked to rate their chances of falling asleep while engaged at 8 different activities, on a 4-point scale: 0 = would never fall asleep; 1=slight chance of falling asleep; 2=moderate chance of falling asleep; 3=high chance of falling asleep. Total score was calculated as the sum of 8 item scores ranging from 0 (never) to 24 (high chance of falling asleep). Higher scores indicate high chances of falling asleep.
Time Frame: Baseline, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 23
units on a scale | 0.7 (3.51)

8. Secondary Outcome: Change From Baseline in the Movement Disorder-Childhood Rating Scale (MD-CRS) Part I Total Score (General Assessment, Centrally Read)
Description: The MD-CRS part I evaluates the impact of dyskinesia in cerebral palsy (DCP) on the activities of the participant and provides a general assessment of the movement disorder of motor function (7 items), oral/verbal function (3 items), self-care (3 items), and attention/alertness (2 items) on a scale of 0 (present) to 4 (absent). All items were scored by the rater in the clinic and were centrally read based on video recording. The total score was obtained by summing the individual items' scores and ranges from 0 (marked/prolonged disorder) to 60 (absent of a disorder), with higher scores indicating lesser disorder.
Time Frame: Baseline, Week 53, Week 54
Population: The ITT analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 30
units on a scale
  Change at Week 53 | -2.41 (5.24)
  Change at Week 54: number analyzed (Participants) | 25
  Change at Week 54 | -1.40 (4.989)

9. Secondary Outcome: Change From Baseline in the MD-CRS Part II Total Score (Movement Disorder Severity, Centrally Read)
Description: MD-CRS part II evaluates the severity of movement disorder on a scale of 0 to 4 in 7 body regions, all areas in which dyskinesia can be seen. All items were scored by the rater in the clinic and were centrally read based on video recording. In rating the movement disorder of a body part, 0 refers to absence of a movement disorder and 4 refers to a situation where movement disorder is present during all of the tasks for the region examined and/or involves 3 or more of the other regions, making completion impossible. The 7 body regions are (i) eye and periorbital region, (ii) face, (iii) tongue and perioral region, (iv) neck, (v) trunk, (vi) upper limb, and (vii) lower limb. Total score was obtained by summing the individual items scores and ranges from 0 (absent of a movement disorder) to 28 (marked/prolonged movement disorder), with higher scores indicating more movement disorder.
Time Frame: Baseline, Week 53, Week 54
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 25
units on a scale
  Change at Week 53 | -1.5 (3.91)
  Change at Week 54: number analyzed (Participants) | 21
  Change at Week 54 | 0.5 (4.34)

10. Secondary Outcome: Change From Baseline in the MD-CRS Part I Total Score (General Assessment, Physician Rated)
Description: The MD-CRS part I evaluates the impact of DCP on the activities of the participant and provides a general assessment of the movement disorder of motor function (7 items), oral/verbal function (3 items), self-care (3 items), and attention/alertness (2 items) on a scale of 0 (present) to 4 (absent). All items were scored by the investigational center physician. The total score was obtained by summing the individual items' scores and ranges from 0 (marked/prolonged movement disorder) to 60 (absent of a movement disorder), with higher scores indicating lesser movement disorder.
Time Frame: Baseline, Week 53, Week 54
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale
  Change at Week 53 | -2.6 (3.70)
  Change at Week 54: number analyzed (Participants) | 24
  Change at Week 54 | -1.4 (3.72)

11. Secondary Outcome: Change From Baseline in the MD-CRS Part II Total Score (General Assessment, Physician Rated)
Description: The MD-CRS part II evaluates the severity of the movement disorder on a scale of 0 to 4 in 7 body regions, all areas in which dyskinesia can be seen in participants with CP. All items were scored by the investigational center physician. In rating the movement disorder of the body part, 0 refers to absence of a movement disorder and 4 refers to a situation where movement disorder is present during all of the tasks for the region examined and/or involves 3 or more of the other regions, making completion impossible. The 7 body regions are (i) eye and periorbital region, (ii) face, (iii) tongue and perioral region, (iv) neck, (v) trunk, (vi) upper limb, and (vii) lower limb. The total score was obtained by summing the individual items' scores and ranges from 0 (absent of a movement disorder) to 28 (marked/prolonged movement disorder), with higher scores indicating more movement disorder.
Time Frame: Baseline, Week 53, Week 54
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale
  Change at Week 53 | -3.12 (4.255)
  Change at Week 54: number analyzed (Participants) | 24
  Change at Week 54 | -1.88 (3.927)

12. Secondary Outcome: Change From Baseline in MD-CRS Global Index Score (Calculated From MD-CRS Parts I and II Total Scores, Physician Rated)
Description: The MD-CRS Global Index is a global measure of the MD-CRS that consolidates the information from parts I and II using the method of weighted means of the 2 normalized indexes obtained from each part. The standardized/normalized score for each item of MD-CRS parts I and II with value X is calculated using the formula: Xst = X - Xmin divided by Xmax - Xmin, where Xmax is the maximum value for the score, and Xmin is the minimum value for the score, or 4 and 0 respectively. The normalized index for the scale, MD-CRS parts I or II, Index I or II, is calculated as the mean value of Xst. The MD-CRS Global Index is the weighted mean of the normalized indexes for centrally read MD-CRS parts I and II using the formula: Global index = n1 * index 1 + n2 * index 2 divided by n1 + n2, where n1 and n2 are the numbers of items in MD-CRS parts I and II respectively. The minimum score is 0 (better) and the maximum score is 1 (worse). The higher score indicates more severe movement disorder.
Time Frame: Baseline, Week 53, Week 54
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale
  Change at Week 53 | -0.1 (0.07)
  Change at Week 54: number analyzed (Participants) | 24
  Change at Week 54 | -0.0 (0.07)

13. Secondary Outcome: Change From Baseline in MD-CRS Global Index Score (Calculated From MD-CRS Parts I and II Total Scores, Centrally Read)
Description: as for outcome 12
Time Frame: Baseline, Week 53, Week 54
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 30
units on a scale
  Change at Week 53 | -0.0 (0.08)
  Change at Week 54: number analyzed (Participants) | 25
  Change at Week 54 | -0.0 (0.06)

14. Secondary Outcome: Change From Baseline in Caregiver Global Impression of Improvement (CaGI-I) Scale Score (Global, Caregiver Rated) at Week 54
Description: The CaGI-I is single item questionnaire to assess the caregiver's impression of improvement in dyskinesia symptoms after initiating therapy. The scale is a caregiver-reported outcome that aims to evaluate all aspects of participants' health and determine if there has been an overall improvement or not in dyskinesia symptoms. The caregiver selected the 1 response from the response options that gave the most accurate description of change in dyskinesia symptoms of the participant they cared for from the beginning of the study: 1=very much improved (since the initiation of treatment); 2=much improved; 3=minimally improved; 4=no change from baseline (symptoms remain essentially unchanged); 5=minimally worse; 6=much worse; 7=very much worse (since the initiation of treatment). The change from baseline CaGI-I score can range from -6 to 6.
Time Frame: Baseline, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 23
units on a scale | -0.6 (1.20)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression of Improvement (CGI-I) Scale Score (Global, Physician Rated) at Week 54
Description: CGI-I is a clinician-reported outcome with a 7-point Likert scale to compare participant's condition to the baseline condition: 1=very much improved since initiation of treatment (nearly all better; good level of functioning; minimal symptoms; represents a very substantial change); 2=much improved (notably better with significant reduction of symptoms; increase in level of functioning but some symptoms remain); 3=minimally improved (slightly better with little or no clinically meaningful reduction of symptoms; represents very little change in basic clinical status, level of care, or functional capacity); 4=no change from baseline (symptoms remain unchanged); 5=minimally worse (slightly worse but may not be clinically meaningful); 6=much worse (clinically significant increase in symptoms and diminished functioning); 7=very much worse since initiation of treatment (severe exacerbation of symptoms and loss of functioning). The change from baseline CGI-I score can range from -6 to 6.
Time Frame: Baseline, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 24
units on a scale | -0.2 (0.88)

16. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Scale Score (Global, Physician Rated) at Week 54
Description: The CGI-S uses a 7-point Likert scale to assess dyskinesia severity as follows (with anchor points for choosing the most appropriate severity level caused by DCP): 1=normal (not at all ill, symptoms of disorder not present past 7 days); 2=borderline (subtle or suspected pathology); 3=mild (clearly established symptoms with minimal, if any, distress or difficulty in social and/or occupational function); 4=moderate (overt symptoms causing noticeable, but modest, functional impairment or distress; symptom level may warrant medication); 5=marked (intrusive symptoms that distinctly impair social/occupational function or cause intrusive levels of distress); 6=severe (disruptive symptoms, behavior, and function are frequently influenced by symptoms, may require assistance from others); 7=extreme (symptoms drastically interfere in many life functions; may be hospitalized). Higher scores indicating more severity.
Time Frame: Baseline, Week 54
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 24
units on a scale | -0.3 (0.64)

17. Secondary Outcome: Change From Baseline in Pediatric Evaluation Disability Inventory-Computer Adapted Test (PEDI-CAT) Score (Activities of Daily Living [ADL], Caregiver Completed, Content-Balanced Version) at Week 53
Description: The PEDI-CAT measures function in 4 domains: (1) Daily Activities; (2) Mobility; (3) Social/Cognitive, and (4) Responsibility. The content-balanced version presents a balance of items from each of the Daily Activities domain's content areas (Getting Dressed, Keeping Clean, Home Tasks, and Eating and Mealtime). A total of approximately 30 items were administered. PEDI-CAT software utilizes Item Response Theory statistical models to estimate a child's abilities from a minimal number of the most relevant items or from a set number of items within each domain. The CAT program then displays the results: normative standard scores, scaled scores, and SE. Scaled score is reported in this endpoint. Scaled scores are based on an estimate of the placement of an individual child along the hierarchical scale within each domain. PEDI-CAT scaled scores are currently on a 20 (lesser improvement) to 80 (more improvement) scale metric. Higher scores indicate greater improvement in functional skills.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 18
units on a scale | 0.9 (2.39)

18. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Chorea (UHDRS-TMC) Score (Centrally Read) at Week 53
Description: The UHDRS-TMC is part of the Unified Huntington's Disease Rating Scale-Total Motor Score (UHDRS-TMS) assessment and assesses the severity of chorea in the 7 body parts: face, mouth, trunk, and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). The central rating was done for all participants, based on the videos collected for the central rating of MD-CRS. The TMC score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 28 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 25
units on a scale | 0.0 (3.20)

19. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Dystonia (UHDRS-TMD) Score (Centrally Read) at Week 53
Description: The UHDRS-TMD is part of the UHDRS-TMS assessment and assesses the severity of dystonia in the 5 body parts: trunk and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). The central rating was done for all participants, based on the videos collected for the central rating of MD-CRS. The TMD score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 20 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 25
units on a scale | -1.0 (3.38)

20. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Motor Score (UHDRS-TMS) Score (Physician Rated) at Week 53
Description: The UHDRS comprises a broad assessment of features associated with Huntington's disease (HD). It is a research tool that has been developed to provide a uniform assessment of the clinical features and course of HD. The Total Motor Score assessment of the UHDRS (UHDRS-TMS) comprises 15 items and assesses eye movements, speech, alternating hand movements, dystonia, chorea, and gait. The UHDRS-TMS was calculated as the sum of the 31 motor assessments; each of which ranged between 0 (absent) to 4 (worst). All items were scored by the investigational center physician. TMS score is a sum of individual scores ranging from 0 (normal motor function) to 124 (severely impaired motor function), with lower scores indicating better motor function.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale | -7.8 (7.78)

21. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Chorea (UHDRS-TMC) Score (Physician Rated) at Week 53
Description: The UHDRS-TMC is part of the UHDRS-TMS assessment and assesses the severity of chorea in the 7 body parts: face, mouth, trunk, and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). All items were scored by the investigational center physician. The TMC score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 28 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale | -3.9 (4.50)

22. Secondary Outcome: Change From Baseline in Unified Huntington's Disease Rating Scale-Total Maximal Dystonia (UHDRS-TMD) Score (Physician Rated) at Week 53
Description: The UHDRS-TMD is part of the UHDRS-TMS assessment and assesses the severity of dystonia in the 5 body parts: trunk and the 4 extremities (right and left upper extremities, right and left lower extremities). Each part was rated from 0 (absent) to 4 (prolonged). All items were scored by the investigational center physician. The TMD score was obtained by adding up each of the separate scores and ranged from 0 (absent) to 20 (marked/prolonged), with higher scores indicating the worse symptoms.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 26
units on a scale | -0.9 (1.65)

23. Secondary Outcome: Change From Baseline in Canadian Occupational Performance Measure (COPM) (Physician Rated) Score at Week 53
Description: The COPM, a semi-structured interview, was used to assess a participant's perception of performance in the areas of self-care, productivity and leisure. The COPM involves a 5-step process within a semi-structured interview conducted by a therapist. The participants were asked to rate 5 most important activities on a 10-point scale for performance and satisfaction, ranging from 1 (not at all able/satisfied) to 10 (able to perform extremely well/ extremely satisfied). Total score is the average of the total performance and satisfaction subscales. Each subscale score is calculated by adding the scores of all activities and then dividing by the number of the activities. The total change from baseline scores can range from -9 to 9. Higher scores indicated very good performance and high satisfaction.
Time Frame: Baseline, Week 53
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEV-50717
Number analyzed (Participants) | 27
units on a scale | 1.4 (1.36)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 55
Description: The ITT analysis set included all enrolled participants, regardless of whether or not a participant took any TEV-50717.
Arm/Group | TEV-50717
All-Cause Mortality (participants affected / at risk) | 1/44
Serious Adverse Events (participants affected / at risk) | 1/44
Other Adverse Events (participants affected / at risk) | 33/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-50717 (N=44)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TEV-50717 (N=44)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 3 (5)
COVID-19 (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 3 (3)
Akathisia (Nervous system disorders) | 3 (4)
Dystonia (Nervous system disorders) | 3 (7)
Headache (Nervous system disorders) | 3 (3)
Somnolence (Nervous system disorders) | 21 (32)
Insomnia (Psychiatric disorders) | 3 (5)

LIMITATIONS AND CAVEATS:
The study was terminated early due to failure of TV50717-CNS-30080 (parent study) to meet the primary efficacy endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04200352/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT04200352/SAP_001.pdf